CLINICAL TRIAL: NCT03617250
Title: The Correlation Between Neutrophil Lymphocyte Ratio and Platelet Lymphocyte Ratio With Disease Activity in Rheumatoid Arthritis
Brief Title: Neutrophil Lymphocyte Ratio and Platelet Lymphocyte Ratio in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Foad, Principal Investigator, Assiut University
Other Study IDs: RHEUMA
Record Dates: First submitted 2018-07-22; First posted 2018-08-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2020-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active patients: 50 rheumatoid patients with active disease according to Disease Activity Score-28
  Interventions: Other: Disease Activity Score-28
- patients with remission: 50 patients with remission according to Disease Activity Score-28
  Interventions: Other: Disease Activity Score-28

INTERVENTIONS:
Other: Disease Activity Score-28 — Assessment of neutrophil-lymphocyte ratio and platelet-lymphocyte ratio and their association with Disease Activity Score-28

SUMMARY:
Rheumatoid arthritis is an autoimmune disease characterized by synovial inflammation and joint destruction that follows a relapsing- remitting course.Disease activity assessment is important for rheumatoid arthritis management .Neutrophil lymphocyte ratio and platelet lymphocyte ratio are associated with inflammatory status and can be used to assess disease activity in rheumatoid arthritis

DETAILED DESCRIPTION:
Rheumatoid arthritis is an autoimmune disease characterized by synovial inflammation and joint destruction that follows a relapsing - remitting course and induce severe disability . Rheumatoid arthritis is an inflammatory disease that causes devastating joint destruction if patients are not appropriately treated. It is characterized by symmetric joint involvement, erosion and deformity in the joints as a result of synovial inflammation .Inflammation is the key determinant and primary underlying mechanism leading to disability and increased mortality in patients with rheumatoid arthritis.Disease activity assessment is important for rheumatoid arthritis management, since it could greatly affect the clinical decision. Current disease activity assessment mainly depend on clinical symptoms, signs and laboratory tests. laboratory Investigations are much preferred due to the advantage of less observer variations.

Therefore assessment of inflammation in rheumatoid arthritis with reliable markers is crucial to predict long term outcome of a particular patient. The most commonly used markers for this purpose are ESR and CRP in daily practice. However both of these markers have some limitations such as reflection of short-term inflammatory activity and low discrimination ability with other superimposed conditions.

Systemic inflammation is associated with changes in circulating blood cells quantity and composition. Normochromic anemia, thrombocytosis, neutrophilia and lymphopenia usually occur with many inflammatory conditions so the features of circulating blood cell components can be used for the assessment of inflammatory activity .

Parameters of hemogram, particularly those including immune system elements are important in the assessment of different diseases and or sign. Immune system elements involve the neutrophils, lymphocytes and platelets that have a role in the control of inflammation, while also undergoing changes secondary to inflammation. Patients with rheumatoid arthritis may be found with increasing platelet counts during active stages of the disease. The counts decrease up on remission of inflammation but detailed role played by platelets remains unobvious .

Platelet count, mean platelet volume (MPV), platelet distribution width (PDW) are three useful indices of platelet function reflecting the platelet production rate. .

Gokmen et al 2016 concluded that MPV and neutrophil lymphocyte ratio (NLR) together with acute phase reactant C.reactive Protein(CRP), erythrocyte sedimentation rate (ESR) can be a useful indices for showing inflammation in RA patients and demonstrated that MPV negatively correlated with CRP and NLR positively correlated with ESR, CRP and anti cyclic citrullinated peptide antibody (antiCCP). The author concluded that high NLR levels in patients with RA is important in predicting prognosis of disease and development of more joint damage and hypothesized that NLR may be Considered to be an indicator of inflammation, disease activity and disease prognosis.

Previous studies have shown that increased neutrophil to lymphocyte ratio (NLR) and platelet to lymphocyte ratio (PLR) are associated with poor prognosis of various inflammatory related diseases such as cancer, chronic kidney disease , acute pancreatitis ) and myocardial infarction . This may be due to the fact that both PLR and NLR are associated with the inflammatory status .

Based on these Studies recently Fu el at., in 2015 hypothesized that both NLR and PLR correlated with the disease activity of RA and suggested that NLR and PLR may be indices for assessment of RA disease activity.

Uslu et al 2015 demonstrated that NLR and PLR were elevated in rheumatoid arthritis patients with active disease compared with patients in remission. So they concluded that NLR and PLR were two new inflammatory markers which could be used to assess disease activity in patients with rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria

* One hundred patients suffering from Rheumatoid arthritis .

Exclusion Criteria:

Patients with:

* Diabetes mellitus, hypertension, acute or chronic renal failure, acute or Chronic liver disease obstructive lung disease, Coronary artery disease.
* Hematologic disorders other than anemia or history of receiving blood transfusion during the past three months.
* Acute or chronic infections.
* Pregnancy or in the postpartum period.
* History of allergic diseases or any malignant disease.
* Patients with leucocytic count less than 4000 u/l

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred rheumatoid arthritis patients divided into two groups. The first group with active disease and the second group with disease remission. There are 50 healthy participants age and sex matched as control group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Assessment of inflammation in rheumatoid arthritis | Average one year
  By using Disease Activity Score-28 to classify patients into patients with active disease and patients with remission

CONTACTS AND LOCATIONS:
Overall Officials: Noha Foad, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Aletaha D, Ward MM, Machold KP, Nell VP, Stamm T, Smolen JS. Remission and active disease in rheumatoid arthritis: defining criteria for disease activity states. Arthritis Rheum. 2005 Sep;52(9):2625-36. doi: 10.1002/art.21235. PMID 16142705
- [Background] Azab B, Jaglall N, Atallah JP, Lamet A, Raja-Surya V, Farah B, Lesser M, Widmann WD. Neutrophil-lymphocyte ratio as a predictor of adverse outcomes of acute pancreatitis. Pancreatology. 2011;11(4):445-52. doi: 10.1159/000331494. Epub 2011 Sep 28. PMID 21968329
- [Background] Briggs C. Quality counts: new parameters in blood cell counting. Int J Lab Hematol. 2009 Jun;31(3):277-97. doi: 10.1111/j.1751-553x.2009.01160.x. PMID 19452619
- [Background] Colglazier CL, Sutej PG. Laboratory testing in the rheumatic diseases: a practical review. South Med J. 2005 Feb;98(2):185-91. doi: 10.1097/01.SMJ.0000153572.22346.E9. PMID 15759949
- [Background] Hobbs KF, Cohen MD. Rheumatoid arthritis disease measurement: a new old idea. Rheumatology (Oxford). 2012 Dec;51 Suppl 6:vi21-7. doi: 10.1093/rheumatology/kes282. PMID 23221583
- [Background] Kisacik B, Tufan A, Kalyoncu U, Karadag O, Akdogan A, Ozturk MA, Kiraz S, Ertenli I, Calguneri M. Mean platelet volume (MPV) as an inflammatory marker in ankylosing spondylitis and rheumatoid arthritis. Joint Bone Spine. 2008 May;75(3):291-4. doi: 10.1016/j.jbspin.2007.06.016. Epub 2008 Apr 9. PMID 18403245
- [Background] Kocyigit I, Eroglu E, Unal A, Sipahioglu MH, Tokgoz B, Oymak O, Utas C. Role of neutrophil/lymphocyte ratio in prediction of disease progression in patients with stage-4 chronic kidney disease. J Nephrol. 2013 Mar-Apr;26(2):358-65. doi: 10.5301/jn.5000152. Epub 2012 May 8. PMID 22573523
- [Background] McInnes IB, Schett G. The pathogenesis of rheumatoid arthritis. N Engl J Med. 2011 Dec 8;365(23):2205-19. doi: 10.1056/NEJMra1004965. No abstract available. PMID 22150039
- [Background] Ugur M, Gul M, Bozbay M, Cicek G, Uyarel H, Koroglu B, Uluganyan M, Aslan S, Tusun E, Surgit O, Akkaya E, Eren M. The relationship between platelet to lymphocyte ratio and the clinical outcomes in ST elevation myocardial infarction underwent primary coronary intervention. Blood Coagul Fibrinolysis. 2014 Dec;25(8):806-11. doi: 10.1097/MBC.0000000000000150. PMID 24911455